CLINICAL TRIAL: NCT00961467
Title: Lenalidomide, Melphalan, Prednisone, and Thalidomide (RMPT) for Relapsed/Refractory Multiple Myeloma
Brief Title: RMPT for Relapsed/Refractory Multiple Myeloma
Acronym: RMPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV MM PI 210
Record Dates: First submitted 2009-08-14; First posted 2009-08-19 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/ refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Melphalan; Prednisone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RMPT (Arm A -thalidomide 50 mg/day) (Experimental)
  Interventions: Drug: Revlimid, Melphalan, Prednisone, Thalidomide
- RMPT (Arm B - thalidomide 100 mg/day) (Experimental)
  Interventions: Drug: Revlimid, Melphalan, Prednisone, Thalidomide

INTERVENTIONS:
Drug: Revlimid, Melphalan, Prednisone, Thalidomide — Thalidomide was administered at 50 mg/day.
  Arms: RMPT (Arm A -thalidomide 50 mg/day)
Drug: Revlimid, Melphalan, Prednisone, Thalidomide — Thalidomide was administered at 100 mg/day.
  Arms: RMPT (Arm B - thalidomide 100 mg/day)

SUMMARY:
After the discovery of melphalan and prednisone (MP), many clinical trials evaluated the efficacy of combination chemotherapy, such as VMCP, VBAP, MOCCA in multiple myeloma (MM) patients, without significant clinical benefit. After 40 years, the combination of MP with thalidomide (MPT) or lenalidomide (MPR) or bortezomib (MPV) have finally and consistently shown additive or synergistic effects.In advanced MM, the combination of melphalan, prednisone and thalidomide induced 12% very good partial response (VGPR) rate, while the combination of melphalan and bortezomib showed 15% near complete remission (nCR) rate. In relapsed patients, the combination of bortezomib with MPT (VMPT) induced 43% VGPR rate. Preliminary results indicate that VMPT may induce a CR rate of around 50% in newly diagnosed patients (unpublished results).In preclinical studies thalidomide showed more anti-angiogenesis activity, while lenalidomide showed more immunomodulatory effects, thus suggesting a combined clinical approach for these two drugs. The toxicity profile of lenalidomide is completely different from that of thalidomide and no cumulative toxicities are expected, again suggesting a combination approach. This study will evaluate the safety and efficacy of combining Lenalidomide, Melphalan, Prednisone and Thalidomide (R-MPT) as salvage treatment for relapsed/refractory myeloma patients. This association might further increase the response rate achieved by the standard oral MPT or MPR regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of a legally consenting age as defined by local regulations.
2. Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
3. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
4. Female patient is either post-menopausal for 24 consecutive months or surgically sterilised or agree to continuous abstinence from heterosexual sexual contact or willing to use two acceptable method of birth control at the same time (one highly effective method and one additional effective method)(Highly Effective Methods: Intrauterine device -IUD-; Hormonal -birth control pills, injections, implants-; tubal ligation; partner's vasectomy; Additional Effective Methods: Latex condom; Diaphragm; Cervical Cap) for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Lenalidomide therapy.
5. Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Lenalidomide therapy.
6. Patient was previously diagnosed with symptomatic multiple myeloma based on standard criteria (12), and has measurable disease, defined as follows:

   * Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours;
   * Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmacytoma > 2cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).
7. Patient is relapsed or refractory after one or two lines of treatment
8. Patient has a Karnofsky performance status ≥ 60%.
9. Patient has a life-expectancy > 3 months.
10. Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):

    * Platelet count ³ 100 x 109/L without transfusion support within 7 days before the test
    * Absolute neutrophil count ³ 1.0 x 109/L without the use of growth factors
    * Total bilirubin £ 1.5 x the ULN
    * AST (SGOT) and ALT (SGPT) £ 2.5 x ULN
    * Corrected serum calcium < 14 mg/dl (3.5 mmol/L)
    * Calculated or measured creatinine clearance: ≥ 20 mL/minute

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or beast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other concomitant standard/experimental anti-myeloma drug or therapy
5. Prior induction therapy with R-MP or M-PT association
6. Any of the following laboratory abnormalities:

   * Platelet count < 100 ´ 109/L.
   * Absolute neutrophil count <1.0 ´ 109/L.
   * Aspartate transaminase (AST): >2.5 x the upper limit of normal (ULN).
   * Alanine transaminase (AST): > 2.5 x the ULN.
   * Total bilirubin: > 1.5 x the ULN.
   * Corrected serum calcium >14 mg/dL (3.5 mmol/L).
   * Calculated or measured creatinine clearance <20 mL/minute
7. Known positive for HIV or active infectious hepatitis, type B or C.
8. Patient has ³Grade 2 peripheral neuropathy within 14 days before enrollment.
9. Known hypersensitivity to thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Myeloma response rate in terms of partial remission (PR) and very good partial remission (VGPR) | 4 years

SECONDARY OUTCOMES:
progression free survival and overall survival | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera S Giovanni Battista, Torino, Italy/Torino, Italy